CLINICAL TRIAL: NCT00155493
Title: Age-Related Changes in Proliferation and Differentiation Capacity of Human Preadipocytes From Periorbital Fat.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 9461700633
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-06

CONDITIONS: Aging

INTERVENTIONS:
Procedure: obtain surgical specimen for analysis

SUMMARY:
Periorbital rejuvenation has been an issue of great interest in plastic surgery. Adipose tissue plays an important role in the periorbital anatomy, and has a great impact on the aging process of the region. We believe age-related atrophy of the facial adipose tissue may be related to the decreased proliferation and differentiation capability of the preadipocytes (adipose precursor cells).

DETAILED DESCRIPTION:
Understanding the age-related changes in periorbital adipose tissue is crucial for improving current rejuvenation techniques, or developing new ones. However, no such study has been reported in the literature.

Hundreds of people came to our hospital requesting upper blepharoplasty every year. Taking advantage of the discarded soft tissue in the blepharoplasty surgery, samples of bilateral pretarsal fat can be easily obtained from patients of various ages. This study is designed to objectively evaluate the age-related changes of the preadipocytes in human periorbital adipose tissue regarding their proliferation and differentiation capability.

The adipose samples taken during the surgery are sent to the lab immediately to separate the preadipocytes from the specimens. Their number is estimated under the microscope, and then the cells are cultured in vitro to evaluate their proliferation and differentiation capability. Proliferation is assessed by counting the number of preadipocyte everyday for 7 days, and differentiation is assessed by Glycerol-3-phosphate dehydrogenase (GPDH) assay.

A linear regression analysis is used to analyze correlations of the parameters with age. Moreover, by dividing the subjects who had their periorbital fat sampled during upper blepharoplasty operation into three age groups, the parameters are compared with ANOVA test. Therefore, the age-related changes of the proliferation and differentiation capability of the preadipocytes in human periorbital adipose tissue can be concluded.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving lower blepharoplasty

Exclusion Criteria:

* patients who do not require fat removal

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-01; Study Completion 2006-08

PRIMARY OUTCOMES:
preadipocyte proportion in aged versus young group

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Bih Tang, M.D. Ph.D., Principal Investigator — National Taiwan University Hospital